CLINICAL TRIAL: NCT06809439
Title: Comparison of Salivary RANKL, OPG, IL-10, IL-1β and Cortisol Levels With Non-surgical Periodontal Treatment in Periodontitis Patients Living in Two Different Geographical Regions in Turkey
Brief Title: Comparison of Saliva Biomarkers in Two Different Geographical Regions of Turkey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Collaborators: Ataturk University (Other); Ankara University (Other)
Responsible Party: Principal Investigator, Sevilay Yeğinoğlu, Asst Prof Dr, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ApprovalNo:11/04, 09.05.2022; TSA-2022-2551 (Other Grant/Funding Number: Ankara University Scientific Research Projects Office)
Record Dates: First submitted 2025-01-16; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-09

CONDITIONS: Saliva; Cortisol; Smoking, Tobacco; Periodontal Bone Loss; Periodontal Disease; Periodontal Therapy
Keywords: RANKL; osteoprotegerin; interleukin-10; non-surgical periodontal therapy; periodontitis; saliva; enviromental; geographical locations
MeSH Terms: conditions — Tobacco Smoking; Alveolar Bone Loss; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: A total of 77 subjects in Ankara and Erzurum, 19 non-smokers (NS-P) with stage III, grade B generalized periodontitis and 14 smokers (SP) with stage III, grade C generalized periodontitis, as well as 22 non-smokers (NS-C) and 22 smokers (SC) periodontally healthy control cases were included in the study.Periodontal parameters were recorded, and unstimulated saliva samples were collected from all patients. Periodontitis patients (N=33) were evaluated clinically and biochemically (saliva IL-1β, cortisol, RANKL, OPG, and IL-10) 4 weeks after complete oral cleansing and root correction (SRP). Saliva samples were analyzed using enzyme-linked immunosorbent assay (ELISA). The data were analyzed using the SPSS software version 22.0.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Ankara (Experimental): Healthy group at Ankara University. Total smokers and non-smokers with clinically healthy gingiva, no deep gingival pockets (≤3mm) and no attachment loss, no bleeding on probing or <10%, no radiographic bone loss were included in the study.
  Clinical parameters were recorded and saliva was collected in this group.
  Interventions: Diagnostic Test: Saliva Collection (Baseline); Other: Probing
- Control Atatürk (Experimental): Healthy group at Atatürk University. A total of patients with clinically healthy gums, no deep gingival pockets (≤3 mm) and attachment loss, no bleeding on probing or <10%, no radiographic bone loss, smokers and non-smokers were included in the study. Clinical parameters were recorded and saliva was collected in this group.
  Interventions: Diagnostic Test: Saliva Collection (Baseline); Other: Probing
- Periodontitis Ankara (Experimental): Smoker patient who applied to Ankara University, Faculty of Dentistry, Department of Periodontics, diagnosed with Stage III periodontitis with a clinically probed pocket depth of more than 5 mm and radiographically ≥3 mm bone loss, smoker patient diagnosed with Stage III.In this group, baseline and post-treatment clinical parameters were recorded and saliva was collected.
  Interventions: Procedure: Non-Surgical Intervention; Diagnostic Test: Saliva Collection (Baseline); Other: Probing; Diagnostic Test: Saliva Collection (After treatment)
- Periodontitis Atatürk (Experimental): Twenty-two patients who applied to the Department of Periodontics, Faculty of Dentistry, Ataturk University, and were diagnosed with Stage III Grade A periodontitis, 11 smokers and 11 smokers, with clinically probed pocket depths greater than 5 mm and radiographically ≥3 mm bone loss.
  Interventions: Procedure: Non-Surgical Intervention; Diagnostic Test: Saliva Collection (Baseline); Other: Probing; Diagnostic Test: Saliva Collection (After treatment)

INTERVENTIONS:
Procedure: Non-Surgical Intervention — Oral hygiene instructions including tooth brushing, flossing, and interdental brushing were given to all patient groups before non-surgical periodontal treatment. In both periodontitis groups, scaling, and root surface smoothing were performed using ultrasonic instruments (Woodpecker Medicals Ins. Co., USA) and Gracey Curettes (Hu-Friedy, Chicago, IL, USA) under local anesthesia once a week for 4 weeks.
  Arms: Periodontitis Ankara; Periodontitis Atatürk
Diagnostic Test: Saliva Collection (Baseline) — Unstimulated saliva samples were collected from all participants between 9:00 and 11:00 am. Clinical periodontal measurements were performed after saliva collection to prevent contamination (bleeding, etc.). Participants refrained from brushing their teeth the morning before sampling and from eating, drinking, or smoking for at least 2 hours before sampling. Patients were asked to rinse their mouths with distilled water 5 minutes before saliva collection. A saliva sample was then collected by spitting directly into a sterile tube. Sample collection was continued for 5 minutes.
Other: Probing — Clinical and radiographic evaluations were performed by trained and calibrated examiners at Ankara University (SY) and Ataturk University (OT). Clinical parameters of probing depth (PPD), clinical attachment level CAL, plaque index PI, and bleeding on probing (BOP) were recorded from six tooth regions (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, middle lingual, and disto-lingual) using periodontal probe. Bone loss was assessed using panoramic radiographs, confirming the diagnosis of periodontitis.
Diagnostic Test: Saliva Collection (After treatment) — Unstimulated saliva samples were collected from all participants between 9:00 and 11:00 am. Clinical periodontal measurements were performed after saliva collection to prevent contamination (bleeding, etc.). Participants refrained from brushing their teeth the morning before sampling and from eating, drinking, or smoking for at least 2 hours before sampling. Patients were asked to rinse their mouths with distilled water 5 minutes before saliva collection. A saliva sample was then collected by spitting directly into a sterile tube. Sample collection was continued for 5 minutes.
  Arms: Periodontitis Ankara; Periodontitis Atatürk

SUMMARY:
Periodontitis is a multifactorial, chronic inflammatory disease caused by many factors such as pathogenic microorganisms, host response, environmental and systemic factors. Immune mechanisms triggered by host-bacteria interaction can initiate tissue destruction by leading to the release of large amounts of inflammatory mediators such as IL-1β. It is thought that IL-10 has a regulatory role by limiting the initiation and progression of the acute inflammatory response with its anti-inflammatory effect. The high detection of RANKL and RANKL/OPG ratios in periodontitis indicates that these markers play a role in bone destruction. Elucidating the connections between the immune system and bone-related cytokines will contribute significantly to the resolution of these complex mechanisms underlying periodontal diseases. Risk factors for periodontal diseases include gender, age, smoking and some hereditary factors. Cortisol is an important marker of psychological stress. It is emphasized that stress and depression reduce immune system function and cause chronic inflammation. Thus, it indirectly provokes periodontal tissue destruction.

DETAILED DESCRIPTION:
This study consists of patients and healthy volunteers. Saliva will be collected only once from healthy volunteers; from patients at the beginning and after non-surgical periodontal treatments are performed by the researchers. In the collected saliva; clinical parameters and salivary RANKL, OPG, IL-10, IL-1β, cortisol levels will be determined in periodontitis and periodontally healthy individuals living in two different geographical regions in Turkey (Ankara -Erzurum); it will be determined whether non-surgical periodontal treatment has an effect on cytokines determined in saliva and clinical status at the end of 1-month follow-up period; periodontal pathogenesis and host response will be evaluated in smoker and non-smoker groups. Analyses will be performed by ELISA method.

The study is based on the hypothesis that "different regional and geographical conditions determining climate, culture, environment, life, stress situations affect the course of periodontitis disease and host response". A regional comparison will be made between markers that affect the course of periodontitis disease and play a role in its pathogenesis in patients with different climate, living and cultural conditions, according to location.

ELIGIBILITY:
Inclusion Criteria:

* 35-60 years of age
* good cooperation
* a minimum of 20 permanent teeth, excluding third molars

Exclusion Criteria:

* systemic diseases
* taking any medications
* received antibiotic treatment in the last three months
* those who had undergone periodontal treatment six months ago
* pregnant or breastfeeding patients
* prosthetic restorations
* undergoing orthodontic treatment

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Study population, pre-treatment and post-treatment periodontal clinical parameters | up to 4 weeks
  This study included 10 systemically healthy non-smokers from Ankara with stage III, grade B generalized periodontitis, 8 smokers with stage III, grade C generalized periodontitis, 11 periodontally healthy non-smokers, and 11 periodontally healthy smokers. In Erzurum, systemically healthy, 9 non-smokers, stage III B generalized periodontitis , 6 smokers (≥10/day), stage III C generalized periodontitis, 11 periodontally healthy non-smokers, and 11 periodontally healthy smokers were included. Clinical parameters of probing depth (PPD), clinical attachment level (CAL), plaque index (PI), and bleeding on probing (BOP) were recorded . All clinical measurements were made after saliva samples were taken and recorded as initial values. The periodontal index form was used for this purpose. (https://www.periodontalchart-online.com/uk/) Nonsurgical periodontal treatments lasted 4 weeks. Baseline and post-treatment periodontal parameters were compared.

SECONDARY OUTCOMES:
Salivary biomarkers | up to 2 months
  Saliva IL-1β (pg/ml), cortisol (ng/ml), RANKL (pg/ml), OPG(ng/ml), and IL-10 (pg/ml) concentrations were assessed via ELISA. The baseline saliva of the control groups and the pre- and post-treatment salivary biochemical parameters of the treatment groups were similar in both cities evaluated.

OTHER OUTCOMES:
Determination of Pocket Depth (PD) | up to 4 weeks
  Williams periodontal probe was used to determine pocket depth. Care was taken to use the probe parallel to the long axis of the tooth with its own weight during the measurements.
  PD was measured from 6 regions (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual/palatal, mid-lingual/palatal, disto-lingual/palatal) for each tooth and recorded in millimeters (mm). The PD value for each tooth was obtained by taking the average of the 6 measured values.
Determination of Clinical Attachment Level (CAL) | up to 4 weeks
  In order to determine CAL, the cementoenamel border will be determined as a reference point and the distance between the reference point and the pocket base will be measured with a periodontal probe and recorded in mm.
  CAL will be recorded from 6 regions (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual/palatal, mid-lingual/palatal, disto-lingual/palatal) for each tooth. The CAL value for each tooth will be obtained by averaging the 6 measured values.
Determination of the Presence and Accumulation Level of Dental Plaque | up to 4 weeks
  Plaque accumulation around the tooth will be recorded using the Plaque Index (PI) developed by Silness and Löe. Accordingly; 0. No plaque,
  1. Presence of plaque in the form of a film attached to the free gingival margin and adjacent tooth surface and detectable with the help of a periodontal probe,
  2. Presence of soft attachment visible to the naked eye at the gingival margin and on the tooth surface,
  3. Presence of extremely soft attachment at the gingival margin and on the tooth surface.
  The PI value of each measured tooth will be obtained by averaging the scores recorded from 4 regions (mid-mesial, mid-buccal, mid-distal, mid-lingual/palatal) for a tooth. The PI value for each patient will be calculated as follows:
  PI= Total PI in all teeth / Total number of teeth
Determination of Gingival Bleeding on Probing | up to 4 weeks
  The Probing Bleeding Index (BPI) developed by Ainamo and Bay will be used to evaluate gingival bleeding on probing.
  According to this index;
  Positive (+) indicates the presence of bleeding on probing,
  negative (-) indicates the absence of bleeding on probing. After applying pressure by the weight of the probe within the pocket using the BPI ; periodontal probe, each tooth will be evaluated for 4 regions (mid-mesial, mid-buccal, mid-distal, mid-lingual/palatal) and will be determined as positive (+) or negative (-) and recorded as a percentage.
  The percentage of bleeding on probing for each patient will be calculated as follows; BOP (bleeding on probing) percentage = number of teeth with bleeding on probing x100 / total number of teeth
RANKL Measurement | up to 2 months
  RANKL concentrations of saliva samples were measured using a commercial ELISA kit (Catalog No: RE3181H, Reed Biotech, Wuhan, China) following the manufacturer's instructions. The measurement range of the kit was 15.63 pg/mL-1000 pg/mL, sensitivity was 9.38 pg/mL, and inter-assay and intra-assay CV (coefficient of variation) values were <10%. Standard solutions in the range of 15.63 pg/mL-1000 pg/mL were prepared, and the results were calculated using a curve graph. The results were given in pg/mL.
OPG Measurement | up to 2 months
  OPG concentrations of saliva samples were measured using a commercial ELISA kit (Catalog No: RE1765H, Reed Biotech, Wuhan, China) following the manufacturer's instructions. The measuring range of the kit was 0.16 ng/mL-10 ng/mL, sensitivity was 0.1 ng/mL, and inter-assay and intra-assay CV (coefficient of variation) values were <10%. Standard solutions were prepared in the range of 0.16 ng/mL-10 ng/mL, and the results were calculated using a curve graph. The results were given in ng/mL.
IL-10 Measurement | up to 2 months
  IL-10 concentrations of saliva samples were measured using a commercial ELISA kit (Catalog No: RE3187H, Reed Biotech, Wuhan, China) following the manufacturer's instructions. The measurement range of the kit was 1.57 pg/mL-100 pg/mL, sensitivity was 0.94 pg/mL, and inter-assay and intra-assay CV (coefficient of variation) values were <10%. Standard solutions were prepared in the range of 1.57 pg/mL-100 pg/mL, and the results were calculated using a curve graph. The results were given in pg/mL.
IL-1β Analysis | up to 2 months
  IL-1β concentrations of saliva samples were measured using a commercial ELISA kit (Catalog No: RE1074H, Reed Biotech, Wuhan, China) and following the manufacturer's instructions. The measurement range of the kit was 7.82 pg/mL-500 pg/mL, sensitivity was 4.69 pg/mL, and inter-assay and intra-assay CV (coefficient of variation) values were <10%. Standard solutions in the range of 7.82 pg/mL-500 pg/mL were prepared, and the results were calculated using a curve graph. The results were given in pg/mL.
Cortisol Analysis | up to 2 months
  Cortisol concentrations of saliva samples were measured using a commercial ELISA kit (Catalog No: RE10109, Reed Biotech, Wuhan, China) and following the manufacturer's instructions. The measuring range of the kit was 0.31 ng/mL-20 ng/mL, sensitivity was 0.9 ng/mL, and inter-assay and intra-assay CV (coefficient of variation) values were <10%. Standard solutions in the range of 0.31 ng/mL-20 ng/mL were prepared, and the results were calculated using a curve graph. The results were given in ng/mL.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - AnkaraUniversity, Ankara
  - Karabuk University, Karabük

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the saliva biomarker statistics of the study as an excel file when requested. Our Turkish study protocol has also received approval (ethics committee decision).
Supporting Information: Study Protocol, SAP
Time Frame: Start date: 2 January, 2023 End date: 2 January, 2028
Access Criteria: They may request the principal investigator to share the data of the study.

REFERENCES:
- [Background] Mengel R, Bacher M, Flores-De-Jacoby L. Interactions between stress, interleukin-1beta, interleukin-6 and cortisol in periodontally diseased patients. J Clin Periodontol. 2002 Nov;29(11):1012-22. doi: 10.1034/j.1600-051x.2002.291106.x. PMID 12472994
- See also: Ethical approval was obtained from this related institution, as it used to be a clinical research board. — https://www.dentistry.ankara.edu.tr/klinik-arastirmalari-etik-kurulu/